CLINICAL TRIAL: NCT00463320
Title: A Placebo-controlled, Randomized, Dose Rising Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Ocular Doses of Pazopanib in Healthy Adult and Elderly Subjects.
Brief Title: A Study To Evaluate The Safety, Tolerability And Pk Of Pazopanib Eye Drops In Healthy Adult And Elderly Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MD7108238
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Macular Degeneration; Age-related Macular Degeneration
Keywords: Age-related macular degeneration (AMD),; vascular endothelial growth factor (VEGF)receptor (VEGFR); choroidal neovascularization,
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pazopanib eye drops and Allergen Refresh Plus eye drops

SUMMARY:
This is a two-part study to evaluate the safety, tolerability and pharmacokinetics of single (Part A) and repeat (Part B) eye drop doses of pazopanib in healthy adult and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age-related macular degeneration patients diagnosed with subfoveal choroidal neovascularization in the study eye, with all of the following characteristics required:

  * central subfield thickness > 300 microns on investigator-determined OCT (inclusive of subretinal fluid);
  * active subfoveal leakage as determined by investigator-determined fluorescein angiography;
  * minimally classic or occult with no classic D8 lesion;
  * lesion size no greater than 12 disc areas;
  * CNV> 50% of lesion area;
  * < 50% of lesion area with blood;
  * ≤ 25% of lesion area with fibrosis.
* Male or female 50 years of age.
* Best-corrected ETDRS visual acuity in the study eye between 80 to 24 letters inclusive (approximately 20/25 to 20/320 or 4/5 to 4/63) at screening.
* A female subject is eligible to participate if she is of non-childbearing potential defined as either pre-menopausal with a documented tubal ligation or hysterectomy, or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases of postmenopausal status a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory.
* Subject is willing and able to return for all study visits, and is willing and able to comply with all protocol requirements and procedures.
* Subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. If the subject is unable to read the consent form due to visual impairment then the consent must be read to the subject verbatim by person administering the consent, a family member or legally acceptable representative. If the subject is unable to provide written informed consent due to visual impairment, then written informed consent on behalf of the subject must be provided by a legally acceptable representative.

(Note: Consent by legally acceptable representative is allowed where this is in accordance with local laws, regulations and ethics committee policy.)

Exclusion criteria:

* Additional eye disease in the study eye that could compromise best corrected visual acuity (i.e. glaucoma with documented visual field loss, clinically significant diabetic retinopathy, ischemic optic neuropathy, or retinitis pigmentosa).
* CNV in the study eye due to other causes unrelated to age-related macular degeneration.
* The presence of retinal angiomatous proliferation (RAP) in the study eye, as determined by the investigator (confirmation by indocyanine green angiography is not required).
* Geographic atrophy involving the center of the fovea in the study eye.
* Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation of the fundus for photographs, fluorescein angiography and OCT.
* Vitreous, subretinal or retinal hemorrhage in the study eye that is unrelated to AMD.
* More than one prior photodynamic therapy (PDT) treatment in the study eye.
* PDT treatment in the study eye < 12 weeks prior to dosing.
* Previous treatment in the study eye with ranibizumab (Lucentis) or bevacizumab (Avastin) without resolution of exudation (intraretinal and subretinal fluid as documented by OCT).
* Use of any treatment, either approved or experimental, for AMD in the study eye within 60 days of first dose of investigational product.
* Intraocular surgery in the study eye within 3 months of dosing.
* Aphakia or total absence of the posterior capsule (Yttrium aluminum garnet (YAG) capsulotomy permitted) in the study eye.
* History of vitrectomy in the study eye.
* Use of topical ocular medications in the study eye within 7 days of first dose of investigational product or expected use of topical ocular medications during the treatment period, with the exception of artificial tears
* Active treatment in the fellow eye, with the exception of preservative-free artificial tears.
* Current use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoxamine, chloroquine/hydroxychloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol).
* Use of systemic steroids (>10 mg prednisone or equivalent/day) within 14 days of first dose.
* An unwillingness to refrain from wearing contact lenses starting from the screening visit, through the follow-up visit
* Medical history or condition:

  * Uncontrolled Diabetes Mellitus, with hemoglobin A1c (HbA1c) > 10%.
  * Myocardial infarction or stroke within 12 months of screening.
  * Active bleeding disorder.
  * Major surgery within 1 month of screening.
  * Hepatic impairment.
* Uncontrolled hypertension, based on criteria provided in Section 7.2.2. Note: Initiation or adjustment of antihypertensive medications is permitted prior to study entry provided the referenced criteria are met.
* ALT or AST above the upper limit of normal or total bilirubin values at or above 1.5 times the upper limit of normal at screening..

Note: Laboratory tests outside of the normal range may be repeated at the discretion of the Investigator.

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result.
* A history of known HIV infection.
* Use of prohibited medications listed in within the restricted timeframe relative to the first dose of study medication.
* History of drug or alcohol abuse within 6 months of the study.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

A condition or situation which, in the opinion of the investigator, may result in significant risk to the patient, confound the study results or interfere significantly with participation.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2007-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Ocular safety by observation and eye exams. | at baseline, each dosing day and follow-up
General safety by PE, VS, cardiac monitoring, clinical laboratory tests and adverse events reporting . | day-1,5,10,14
Pazopanib exposure by AUC and Cmax . | day 1,14

SECONDARY OUTCOMES:
Pazopanib exposure measured by secondary pharmacokinetic parameters at day 1 and 14.
Safety endpoints include complete ophthalmic examination, vital signs (heart rate and blood pressure), cardiac monitoring (electrocardiogram), clinical laboratory tests, clinical monitoring and adverse event reporting.
Change in visual acuity (number of letters read on standardized ETDRS charts).
Change in retinal morphology (i.e. CNV, intraretinal cysts, intraretinal fluid, subretinal fluid, and retinal pigment epithelial detachment) as determined by OCT.
Change in neovascular size, lesion size and characteristics (fibrosis, atrophy, blood) as measured by fluorescein angiography and fundus photography.
Cmax, tmax, and AUC(0-24) of plasma pazopanib, if data are sufficient.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Austin, Texas